CLINICAL TRIAL: NCT00607217
Title: Controlled Trial of Serologic and Clinical Efficacy of Influenza Vaccine in Post-Myocardial Infarction Patients and in Those With Stable Angina Pectoris
Brief Title: The Efficacy of Influenza Vaccination in Patients With Coronary Artery Diseases
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Maryam Keshtkar-Jahromi, Infectious Diseases and Tropical Medicine Research Center, SBMU, Tehran, Iran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SBMU- 86-03-105-5433B; SMMC- 13861008B
Record Dates: First submitted 2008-01-10; First posted 2008-02-05 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2008-09

CONDITIONS: Coronary Artery Diseases; Myocardial Infarction; Stable Angina
Keywords: Coronary artery diseases; Myocardial infarction; Stable angina; Influenza; Vaccine
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Angina, Stable; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CAD-Exp (Experimental): Enrolled coronary artery disease patients who are randomly assigned to receive influenza vaccine
  Interventions: Biological: influenza vaccine
- CAD-Control (Placebo Comparator): Enrolled coronary artery disease patients who are randomly assigned to receive placebo of influenza vaccine
  Interventions: Biological: placebo for influenza vaccine
- Healthy-Control (Experimental): Enrolled healthy subjects serve as control for CAD-Exp
  Interventions: Biological: influenza vaccine

INTERVENTIONS:
Biological: influenza vaccine — Intramuscular injection of one 0.5-mL dose of influenza vaccine
  Other Names: 2006-2007 vaccination campaign of Influvac (SolvayPharma)
  Arms: CAD-Exp
Biological: placebo for influenza vaccine — Intramuscular injection of one 0.5-mL dose of placebo for influenza vaccine
  Arms: CAD-Control
Biological: influenza vaccine — Intramuscular injection of one 0.5-mL dose of influenza vaccine
  Other Names: 2006-2007 vaccination campaign of Influvac (SolvayPharma)
  Arms: Healthy-Control

SUMMARY:
This study wishes to understand:

1. whether vaccination against influenza in coronary artery disease (myocardial infarction and stable angina) patients is as effective as it is in healthy subjects;
2. whether vaccination really decreases the episodes of influenza infection in those coronary artery disease patients who receive the vaccine than those who do not.

DETAILED DESCRIPTION:
Influenza infection may become complicated in patients with chronic conditions, including coronary artery disease (CAD) [1]. Influenza vaccination is now recommended as part of comprehensive secondary prevention in individuals with coronary and other atherosclerotic vascular disease (evidence level: Class I, Level B) [2]. Although there is controversial evidence pro [3,4] and against [5] the efficacy of influenza vaccination in protecting CAD population against cardiovascular events, the efficacy of vaccine in actual reduction in episodes of influenza infection and its fatal complications in CAD patients has not been, to our knowledge, well studied before. Furthermore, we found no report comparing serologic response to the influenza vaccine antigens between CAD patients and healthy controls.

This study aims to identify the efficacy of influenza vaccination in CAD individuals in terms of both serologic response (as compared with healthy individuals) and clinical outcomes (as compared with CAD patients not vaccinated).

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease (CAD) group (CAD-Exp and CAD-Control):
* Patients with the diagnosis of acute, evolving or recent MI (after recovered the acute phase) as defined by:

  1. Typical rise and gradual fall (troponin) or more rapid rise and fall (CK-MB) of biochemical markers of myocardial necrosis with at least one of the following:
* Ischemic symptoms
* Development of pathologic Qwaves on the ECG
* ECG changes indicative of ischemia (ST segment elevation or depression); OR
* Coronary artery intervention (e.g., coronary angioplasty). 2. Pathologic findings of an acute MI [1]:
* Patients with stable angina pectoris (SA) and documented coronary artery stenosis (angiography).
* Healthy Control group: healthy controls, proportionally matched by gender and age with the patient group (separate control groups for MI and SA patients).

Exclusion Criteria:

* Any acute disease
* Chronic liver or kidney diseases
* Conditions accompanied by immunosuppression (like organ transplantation, HIV)
* Diagnosed malignancy
* Incubation with influenza vaccine within the past 5 years
* Any psychological disease that interferes with regular follow-up
* Congestive heart failure (Killip class IV)
* Unstable angina; AND
* Contradictions of vaccine incubation (like egg allergy).

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Influenza infection | 6 months
Serologic response (≥4-fold HI titer rise) to each of the 3 antigens of the trivalent vaccine of the 2006-07 campaign [Solomon Islands/3/2006(H1N1), Wisconsin/67/2005 (H3N2), and Malaysia/2506/2004 - like strains] | 1 month

SECONDARY OUTCOMES:
Magnitude of change in the antibody titer against each of the three influenza vaccine antigens | 1 month
Protective antibody (≥1:40) titer after vaccination | 1 month
Influenza-related death | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Keshtkar-Jahromi, M.D.; M.P.H., Study Chair — Infectious Diseases and Tropical Medicine Research Center, Shaheed Beheshti Medical University, Tehran, Iran; Hossein Vakili, M.D., Principal Investigator — Cardiovascular Research Center, Shaheed Beheshti Medical University, Tehran, Iran; Mohammad Rahnavardi, M.D., Principal Investigator — Infectious Diseases and Tropical Medicine Research Center, Shaheed Beheshti Medical University, Tehran, Iran; Ali Eskandari, MD, Principal Investigator — Shaheed Beheshti University (MC); Sharareh Gholamin, MD, Principal Investigator — Shaheed Beheshti University (MC); Seyed Mostafa Razavi, MD, Principal Investigator — Shaheed Beheshti University (MC)
Locations (1):
- Shaheed Modarres Medical Center, Tehran, Tehran Province, Iran

REFERENCES:
- [Background] Thompson WW, Shay DK, Weintraub E, Brammer L, Bridges CB, Cox NJ, Fukuda K. Influenza-associated hospitalizations in the United States. JAMA. 2004 Sep 15;292(11):1333-40. doi: 10.1001/jama.292.11.1333. PMID 15367555
- [Background] Smith SC Jr, Allen J, Blair SN, Bonow RO, Brass LM, Fonarow GC, Grundy SM, Hiratzka L, Jones D, Krumholz HM, Mosca L, Pasternak RC, Pearson T, Pfeffer MA, Taubert KA; AHA/ACC; National Heart, Lung, and Blood Institute. AHA/ACC guidelines for secondary prevention for patients with coronary and other atherosclerotic vascular disease: 2006 update: endorsed by the National Heart, Lung, and Blood Institute. Circulation. 2006 May 16;113(19):2363-72. doi: 10.1161/CIRCULATIONAHA.106.174516. No abstract available. PMID 16702489
- [Background] Gurfinkel EP, de la Fuente RL, Mendiz O, Mautner B. Influenza vaccine pilot study in acute coronary syndromes and planned percutaneous coronary interventions: the FLU Vaccination Acute Coronary Syndromes (FLUVACS) Study. Circulation. 2002 May 7;105(18):2143-7. doi: 10.1161/01.cir.0000016182.85461.f4. PMID 11994246
- [Background] Leon de la Fuente R, Gurfinkel EP, Toledo D, Mautner B; Grupo de Estudio FLUVACS. [Flu vaccination in patients with acute coronary syndromes: treatment benefit in prespecified subgroups]. Rev Esp Cardiol. 2003 Oct;56(10):949-54. doi: 10.1016/s0300-8932(03)76991-7. Spanish. PMID 14563288
- [Background] Jackson LA, Yu O, Heckbert SR, Psaty BM, Malais D, Barlow WE, Thompson WW; Vaccine Safety Datalink Study Group. Influenza vaccination is not associated with a reduction in the risk of recurrent coronary events. Am J Epidemiol. 2002 Oct 1;156(7):634-40. doi: 10.1093/aje/kwf073. PMID 12244032
- [Background] Alpert JS, Thygesen K, Antman E, Bassand JP. Myocardial infarction redefined--a consensus document of The Joint European Society of Cardiology/American College of Cardiology Committee for the redefinition of myocardial infarction. J Am Coll Cardiol. 2000 Sep;36(3):959-69. doi: 10.1016/s0735-1097(00)00804-4. PMID 10987628